CLINICAL TRIAL: NCT00719979
Title: Integrated Telemental Health Intervention for Depression in Primary Care
Brief Title: Effectiveness of a Technology Assisted Behavioral Intervention in Assisting People With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH078922 (NIH); DSIR 83-ATP (Other Grant/Funding Number: NCT00719979); 5P20MH090318-02 (NIH)
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2013-01

CONDITIONS: Depression
Keywords: Major Depressive Disorder; Cognitive Behavior Therapy; Technology Assisted; Internet; Primary Care
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iCBT and TeleCoaching (Experimental): Participants received the technology-assisted behavioral intervention (iCBT + TeleCoaching).
  Interventions: Behavioral: Behavioral intervention (iCBT + TeleCoach)
- iCBT(MoodManager) (Experimental): Participants received Internet-based cognitive behavioral therapy only.
  Interventions: Behavioral: Behavioral intervention (iCBT + TeleCoach); Behavioral: Internet-based cognitive behavioral therapy (I-CBT)
- Treatment as usual / Wait-list control (Active Comparator): Participants received treatment as usual . For wait-list control, participants were not provided any intervention for 6 weeks, after which they were allowed to choose coached or self-directed moodManager.
  Interventions: Behavioral: Treatment as usual / Wait-list control

INTERVENTIONS:
Behavioral: Behavioral intervention (iCBT + TeleCoach) — TABI will include 12 weeks of Internet-based cognitive behavioral therapy (iCBT) combined with brief telephone and email support from a coach.
  Arms: iCBT and TeleCoaching; iCBT(MoodManager)
Behavioral: Internet-based cognitive behavioral therapy (I-CBT) — I-CBT will include access to an interactive Web-based intervention designed to teach and facilitate the use of cognitive behavioral skills. The intervention will last 12 weeks.
  Arms: iCBT(MoodManager)
Behavioral: Treatment as usual / Wait-list control — TAU will include standard treatment from participants' primary care physicians. Participants will be able to choose between TABI and I-CBT treatment options after a 6-week wait-list period.
  Arms: Treatment as usual / Wait-list control

SUMMARY:
This study will develop and evaluate the effectiveness of a technology-assisted behavioral intervention, consisting of Internet-based cognitive behavioral therapy combined with telephone and email support, in reducing depressive symptoms and improving treatment adherence in primary care patients with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common mental disorder, with up to 10.3% of the population experiencing the disorder in a given 12-month period. Symptoms of MDD include feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; excessive irritability and restlessness; inability to concentrate; and lack of enjoyment in previously enjoyed activities. Fortunately, MDD is treatable with forms of psychotherapy and/or antidepressant medications. Several studies have found that when given a choice, about two-thirds of depressed patients prefer psychotherapy treatment over antidepressant medication. Although psychotherapy treatments are both effective and desirable, a variety of barriers exist to initiating and sustaining psychotherapy. Only about 20% of all patients referred for psychotherapy treatments ever follow up. Of those who do initiate psychotherapy, nearly half drop out before completing treatment.

Delivering an intervention through telecommunication technologies, such as the telephone and Internet, has the potential to overcome many of the barriers to existing treatments for depression. For example, telephone- and Web-based interventions can reduce cost, extend specialized treatment over broad geographic areas, and permit considerable flexibility in scheduling of treatment components. Technology-assisted Behavioral Intervention(TABI) is a specific form of a telecommunication behavioral intervention that incorporates Web-based Internet, e-mail, and telephone intervention. Further study is needed to determine the effectiveness of TABI in reducing depressive symptoms and attrition rates in people with MDD. This pilot study will first develop TABI, which will consist of Internet-based cognitive behavioral therapy (I-CBT) accompanied by telephone and e-mail support. The study will then compare the effectiveness of TABI with the effectiveness of I-CBT alone and treatment as usual (TAU) in reducing depressive symptoms and improving treatment adherence in primary care patients with MDD.

Participation in the treatment phase of this study will last 12 weeks. All participants will first undergo initial assessments that will include a telephone interview and a series of questionnaires about mood. Eligible participants will then be assigned randomly to receive TABI, I-CBT alone, or TAU. Participants assigned to TABI and I-CBT will both undergo 12 weeks of a Web-based Internet intervention consisting of modules to help them learn skills to manage their moods. Participants assigned to TAU will receive standard treatment from their primary care physicians and will be able to choose between TABI and I-CBT treatment options after a 6-week wait-list period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders-IV diagnosis of MDD as assessed using the Mini Mental State Exam (MINI)
* Has a telephone, email account, computer, and broadband access to the Internet
* Able to navigate the Internet
* Able to speak and read English

Exclusion Criteria:

* Hearing or voice impairment
* Visual impairment that would prevent use of the workbook and completion of assessment materials
* Meets criteria for dementia
* Diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance abuse, or other diagnosis for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous
* Currently receiving individual psychotherapy or planning to receive psychotherapy during the 12-week treatment phase of the study
* Planning to be out of town or unavailable for treatment for 4 weeks or more during the scheduled treatment time
* Exhibits severe suicidality, including ideation, plan, and intent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at baseline and Weeks 6 & 12 (post treatment)
  PhQ-9 and diagnosis (using MINI)
Utilization and Attrition | Baseline-Week 12
  # logins

SECONDARY OUTCOMES:
Patient Satisfaction (Satisfaction Index-Mental Health) | Measured at baseline and Weeks 6 & 12

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Mohr DC, Duffecy J, Ho J, Kwasny M, Cai X, Burns MN, Begale M. A randomized controlled trial evaluating a manualized TeleCoaching protocol for improving adherence to a web-based intervention for the treatment of depression. PLoS One. 2013 Aug 21;8(8):e70086. doi: 10.1371/journal.pone.0070086. eCollection 2013. PMID 23990896